CLINICAL TRIAL: NCT07293611
Title: Prospective, Multicenter, Single-arm, Open-label Study to Assess the Safety and Feasibility of the Levita Magnetic Surgical System for Reduced Port in Upper Gastrointestinal Laparoscopic Procedures
Brief Title: A Study at Multiple Centers to Evaluate the Safety and Practicality of the Levita Magnetic Surgical System for Use in Laparoscopic Upper Gastrointestinal Surgeries.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Levita Magnetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LVT011
Record Dates: First submitted 2025-12-12; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Upper Gastrointestinal Laparoscopic Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Magnetic Surgical System in laparoscopic upper gastrointestinal procedures (Experimental)
  Interventions: Device: Levita Magnetic Surgical System

INTERVENTIONS:
Device: Levita Magnetic Surgical System — The Magnetic Surgical System (MSS), which was cleared for market in the U.S. most recently per 510(k) K252435 and is commercially available in Chile, is composed of two hand-held instruments: a Magnetic Grasper and an external Magnetic Controller.
  The Magnetic Grasper is comprised of two main components: a detachable Grasper Tip and a Shaft. The detachable Grasper Tip provided with the Magnetic Grasper is 6.5cm in length. An optional 12.5cm length detachable Grasper Tip may be used as a replacement for the 6.5cm Grasper Tip and can be used with the Shaft interchangeably. The Magnetic Controller is a single unit with handles that is held external to the body and emits a magnetic field that attracts the detachable Grasper Tip.
  In this study the 6.5 Grasper Tip will be used.

SUMMARY:
A Study at Multiple Centers to Evaluate the Safety and Practicality of the Levita Magnetic Surgical System for Use in Laparoscopic Upper Gastrointestinal Surgeries.

ELIGIBILITY:
Inclusion Criteria:

* BMI range of 20 to 60kg/m2
* Scheduled to undergo laparoscopic procedures
* Willing and able to provide a written Informed Consent Form (ICF) to participate in the study prior to any study- required procedures

Exclusion Criteria:

* Individuals with pacemakers, defibrillators, or other electromedical implants
* Individuals with ferromagnetic implants
* American Society of Anesthesiologists (ASA) score of III or IV
* Significant comorbidities: cardiovascular, neuromuscular, chronic obstructive pulmonary disease, and urological disease (renal failure)
* Clinical history of impaired coagulation confirmed by abnormal blood tests
* Individuals who have signs of hepatic abnormality (e.g.: cirrhosis, liver failure, increase in liver enzymes, etc.)
* Anatomical abnormality or disease of intended target tissue noted after initiation of index procedure that would prevent device use
* Pregnant or wishes to become pregnant during the length of study participation
* Individual is not likely to comply with the follow-up evaluation schedule
* Participating in a clinical trial of another investigational drug or device
* Prisoner or under incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Device and/or Procedure Related Adverse Events | From enrollment to end of follow up at 30 days.
  Adverse events will be summarized by relatedness to the device and/or procedure, seriousness and level of severity.
Average Number of Ports | During index procedure.
  Ability to adequately retract the stomach, omentum, and small bowel to achieve effective exposure of the target tissue. Adequate retraction will be deemed to be achieved if an additional port that is typically used for retraction and exposure of target tissues can be eliminated.

CONTACTS AND LOCATIONS:
Locations (2):
- Chile (2):
  - Clinica Colonial, Huechuraba, Santiago Metropolitan
  - Hospital Luis Tisne, Peñalolén, Santiago Metropolitan

IPD SHARING:
Plan to Share IPD: Undecided